CLINICAL TRIAL: NCT05323760
Title: Functional Capacity in Patients Who Recovered From Mild COVID-19 With Exertional Dyspnea.
Brief Title: Functional Capacity in Patients Post Mild COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0760-20-RMB
Record Dates: First submitted 2022-04-07; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: Cardiopulmonary Exercise Testing; COVID-19; Exertional dyspnea
MeSH Terms: conditions — COVID-19 | interventions — Exercise Test

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiopulmonary exercise test (CPET) (Experimental): Cardiopulmonary exercise testing (CPET) using a Quark CPET metabolic cart (Rome, Italy) according to American Thoracic Society (ATS) guidelines. A symptom-limited test on a treadmill will be performed, using incremental ramp Bruce protocol up to exhaustion. Patients who will not be able to perform the test on a treadmill will be tested on a cycle ergometer beginning with a no-resistance warm-up lasting 2-3 minutes, followed by incrementing resistance (8-30 Watts/minute) adapted to the patient's functional capacities according to the examiner's free judgment, up to exhaustion.
  Interventions: Device: Cardiopulmonary exercise test (CPET)

INTERVENTIONS:
Device: Cardiopulmonary exercise test (CPET) — A symptom-limited test on a treadmill will be performed, using incremental ramp Bruce protocol up to exhaustion. Patients who will not be able to perform the test on a treadmill will be tested on a cycle ergometer beginning with a no-resistance warm-up lasting 2-3 minutes, followed by incrementing resistance (8-30 Watts/minute).

SUMMARY:
Patients recovered from mild coronavirus 2019 (COVID-19) disease without pulmonary involvement may experience long-term physical impairment and dyspnea. The investigators aim to characterize physiologic limitations in patients who recovered from mild COVID-19.

Methods: Pulmonary function tests (PFTs), 6-minute walk test (6MWT), echocardiography and cardiopulmonary exercise test (CPET) will be completed in patients recovered from mild COVID-19 disease with prolonged dyspnea (Subgroup "A") and compared to patients recovered from moderate/severe COVID-19 (subgroup "B") and to non-COVID-19 patients with unexplained dyspnea (subgroup "C").

DETAILED DESCRIPTION:
Infection with severe acute respiratory syndrome coronavirus-2 leads to severe disease requiring hospitalization in 20% of the cases. Respiratory failure from severe acute respiratory syndrome coronavirus-2 infection can range from mild pneumonia and hypoxia to life threatening hypoxia secondary to severe acute respiratory distress syndrome requiring intensive care unit and mechanical ventilation in about 12-24% of the hospitalized patients. Most patients are discharged with minimal or no long-term oxygen therapy while others are discharged with ongoing respiratory symptoms and long-term oxygen therapy. In the longer term, there is a significant concern that severe coronavirus disease 2019 can lead to organizing pneumonia and severe acute lung injury with evolution to widespread fibrotic changes as seen in fatal cases of coronavirus disease showing pulmonary fibrosis at autopsy. Studies in severe acute respiratory syndrome survivors, another corona virus infection, showed persistent and significant impairment of exercise capacity and health status over 24 months based on PFTs, 6-minute walk test and health questionnaire. Infection with respiratory syndrome coronavirus-2 has been also associated with multiple direct and indirect cardiovascular complications including acute myocardial injury, myocarditis, arrhythmias, and venous thromboembolism. However, long term cardiovascular consequences from coronavirus disease 2019 are still unknown. The investigators sought to determine the pulmonary, cardiac and other physiologic limitations in patients who recovered from severe coronavirus disease 2019 with physiologic tests including PFTs, echocardiography and cardio-pulmonary exercise test which is currently the most comprehensive physiologic test that can differentiate between the different limitations and add novel data regarding short and long term physiologic consequences of coronavirus disease 2019.

ELIGIBILITY:
Inclusion Criteria:

* Patients recovering from COVID-19 with a documented infection with severe acute respiratory syndrome coronavirus-2 and cognitive ability to sign informed consent and physical ability to participate in exercise tests.

Exclusion Criteria:

* Patients with severe pulmonary, cardiac disease prior to COVID-19, pregnant women, and patients with active infection or cancer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | Measured continuously during 15 minutes of the exercise test (CPET)
  Oxygen uptake evaluated by cardiopulmonary exercise testing (CPET)

SECONDARY OUTCOMES:
Echocardiography | Ten minutes
  Left ventricle shortening and ejection fraction, as well as possible cardiac structural or hemodynamic abnormalities will be evaluated by trans-thoracic echocardiography (iE33, Philips).
Six minute walk test | Six minutes of evaluation, completed pre cardiopulmonary exercise test.
  The distance gained after six minute of habitual walking.
Spirometry | Five minutes before and after the cardiopulmonary exercise testing
  Pulmonary function as assessed by spirometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel